CLINICAL TRIAL: NCT02472600
Title: A Randomized Controlled Multicenter Trial of a Five Day Course of Oral Colistin and Neomycin Followed by Restoration of the Gut Microbiota Using Fecal Transplantation to Eradicate Intestinal Carriage of Extended Spectrum Beta-lactamase or Carbapenemase-producing Enterobacteriaceae in High-risk Patients
Brief Title: Eradication of Antibiotic-resistant Bacteria Through Antibiotics and Fecal Bacteriotherapy
Acronym: R-GNOSIS WP3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stephen Harbarth (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor-Investigator, Stephen Harbarth, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-266; 2014-003727-22 (EudraCT Number)
Record Dates: First submitted 2015-06-04; First posted 2015-06-16 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Intestinal Colonization With Multidrug-resistant Bacteria
Keywords: extended spectrum beta-lactamase producing enterobacteriaceae; carbapenemase producing enterobacteriaceae; multidrug resistant bacteria
MeSH Terms: interventions — Colistin; Neomycin; Fecal Microbiota Transplantation; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- colistin + neomycin followed by FMT (Active Comparator): CAPSULE APPROACH:
  Treatment days 1-5
  * Colistin sulphate 2 million IU per os 4x/day (for 5 days)
  * Neomycin sulphate 500 mg (salt) per os 4x/day (for 5 days) Treatment day 6: no treatment
  Treatment days 7 and 8:
  -15 capsules of capsulized Fecal microbiota transplantation (FMT) per os per day
  NASOGASTRIC TUBE APPROACH:
  Treatment days 1-5
  * Colistin sulphate 2 million IU per os 4x/day (for 5 days)
  * Neomycin sulphate 500 mg (salt) per os 4x/day (for 5 days)
  Treatment day 6 and 7:
  - Omeprazole 20 mg per os 1 dose on the evening of day 6 and on the morning of day 7
  Treatment day 7:
  - Infusion of 80 ml of a standardized stool suspension through a nasogastric tube - Fecal microbiota transplantation (FMT)
  Interventions: Drug: Colistin; Drug: Neomycin; Drug: Fecal microbiota transplantation (FMT); Drug: Omeprazole
- No intervention (No Intervention): Control arm without any intervention

INTERVENTIONS:
Drug: Colistin
  Other Names: Polymyxin E; Diarönt® mono; A07AA10
  Arms: colistin + neomycin followed by FMT
Drug: Neomycin
  Other Names: Neomycin Sulfate X-Gen; A01AB08
  Arms: colistin + neomycin followed by FMT
Drug: Fecal microbiota transplantation (FMT) — FMT consist in the administration of fecal material obtained from healthy donors that has been diluted, homogenized, filtered and reconcentrated. In this study the processed fecal material will be frozen at -80°C after processing and will be administered to patients for up to six months after freezing via a nasogastric tube or via capsules.
  Other Names: Fecal bacteriotherapy; Feces transplantation
  Arms: colistin + neomycin followed by FMT
Drug: Omeprazole — Administered to inhibit gastric acid secretion before FMT administration if FMT administered via nasogastric tube approach (not used for capsule approach).
  Other Names: A02BC01
  Arms: colistin + neomycin followed by FMT

SUMMARY:
This investigator initiated,international, multicenter open-label, randomized controlled trial aims to assess whether a 5 day course of oral nonabsorbable antibiotics (colistin sulfate 2 million IU per os 4x/day and neomycin sulfate 500 mg (salt) per os 4x/day ) followed by fecal microbiota transplantation (administered either via nasogastric administration or via capsules) is effective at eradicating intestinal carriage of beta-lactamase producing Enterobacteriaceae (ESBL-E) and carbapenemase producing Enterobacteriaceae (CPE). compared to no intervention (current standard of care) in adult non-immunosuppressed patients .

DETAILED DESCRIPTION:
In recent years a certain family of bacteria (Enterobacteriaceae) that colonizes the human gastrointestinal tract but can also cause severe infections has increasingly become resistant to antibiotics by acquiring enzymes that can inactivate a wide array of these valuable drugs. Depending on the class of beta-lactam antibiotics that these enzymes can inactivate, these bacteria are either designated as extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E) or carbapenemase producing Enterobacteriaceae (CPE).

The R-GNOSIS project which is financed by the European Commission combines five separate international clinical studies (work packages 2 to 6) that examine intervention strategies to reduce carriage, infection and spread of these bacteria. This study (work package 3 of R-GNOSIS) will be conducted in 4 centers in 3 European countries (Switzerland, France, The Netherlands) and Israel. The study will examine whether it is possible to eradicate intestinal carriage with ESBL-E and CPE by administering a 5 day course of oral nonabsorbable antibiotics (colistin sulfate and neomycin sulfate) followed by administration of "healthy" stool flora obtained from a healthy volunteer donor ("fecal microbiota transplantation" or FMT). The "healthy" stool flora for this procedure will be obtained from carefully selected healthy volunteers that have been tested for a wide variety of infectious diseases and do not show any risk factors or risky behavior for transmittable diseases. Once the fecal material has been processed it will be frozen at -80°C for up to six months until administration to patients (via capsules or via a nasogastric tube). FMT has been successfully used to treat recurrent infections with a specific pathogen (Clostridium difficile) and has proven safe and effective for this indication but has never been studied with the aim of eradicating multidrug-resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years at date of inclusion)
* Ability to provide informed consent
* Documented intestinal carriage of ESBL-E and / or CPE by stool culture at baseline (visit 0)
* IF COLONIZED WITH ESBL-E ONLY (WITHOUT CPE): At least one episode of symptomatic infection with ESBL-E requiring systemic antibiotic therapy within the last 180 days before date of inclusion (based on the last day of antibiotic therapy for that infection)

Exclusion Criteria:

* Pregnancy or planned pregnancy
* Breastfeeding
* Difficult / impossible follow-up
* Allergy or other contraindication to one of the study drugs
* Recurrent aspirations / chronic dysphagia
* Resistance to colistin (defined as MIC> 2 mg/l) of any of the ESBL-E or CPE strains isolated at baseline
* Estimated life expectancy < 6 months
* Treatment with any systemic antibiotic on the day of inclusion
* Severe immunodeficiency

  * Systemic chemotherapy ≤30 days from baseline or planned chemotherapy within the next 6 months
  * Human Immunodeficiency Virus (HIV) with CD4 count < 250/mcl
  * Prolonged use of steroids (prednisone equivalent ≥ 60 mg per day for >= 30 days) or other immunosuppressive medications
  * neutropenia with absolute neutrophil count <1000/μL,
  * Solid organ transplant
  * Hematopoeitic stem cell transplant recipients
  * Other causes of severe immunodeficiency
* Current hospitalization in an Intensive Care Unit
* Estimated glomerular filtration rate (CKD-EPI) < 15 ml/min/1.73m2
* Severe food allergy (anaphylaxis, urticaria)
* Unavailability of compatible FMT preparation (with regard to donor / recipient cytomegalovirus, Epstein-Barr virus and toxoplasma serology)
* Anatomic contraindication to the placement of a nasogastric tube (only if FMT application via nasogastric tube)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11-29 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Intestinal carriage of ESBL-E / CRE | 35 to 48 days after randomization
  Intestinal carriage of ESBL-E / CRE (absence / presence by stool culture of any ESBL-E and / or CRE with enrichment independent of type of carriage at baseline) 35 to 48 days after randomization

SECONDARY OUTCOMES:
Intestinal carriage of ESBL-E / CRE | 6 months after randomization
  Intestinal ESBL-E or CRE carriage (detected / not detected) by stool culture during the other follow-up visits
Occurrence of any adverse drug reaction | 6 months
Occurrence of any adverse event | 6 months
Occurrence of any serious adverse event | 6 months
Occurrence of any gastrointestinal adverse event | 6 months
Isolation of any not intrinsically colistin resistant strain of Enterobacteriaceae during follow-up (MIC> 2mg/l) | 6 months
Comparison between treatment groups of the change (relative to baseline) in the proportion of bacterial taxa and antibiotic resistance genes over time | 6 months
Comparison of the global microbiota composition and diversity between the groups with FMT from the same donor and the groups with FMT from different donors | 6 months
Assess the stability of the microbiome of donor stools after 3 months of frozen storage | 3 months of freezing (donor stools)
  Aliquots from a random sample of donations will also be taken for metagenomic analysis performed after 3 months of storage at -80°C to assess the long-term impact of freezing on the microbiome
Assess the stability of the microbiome of donor stools after 6 months of frozen storage | 6 months of freezing (donor stools)
  Aliquots from a random sample of donations will also be taken for metagenomic analysis performed after 6 months of storage at -80°C to assess the long-term impact of freezing on the microbiome
Assess the stability of the microbiome of donor stools after 12 months of frozen storage | 12 months of freezing (donor stools)
  Aliquots from a random sample of donations will also be taken for metagenomic analysis performed after 12 months of storage at -80°C to assess the long-term impact of freezing on the microbiome
Assess the stability of the microbiome of donor stools after 18 months of frozen storage | 18 months of freezing (donor stools)
  Aliquots from a random sample of donations will also be taken for metagenomic analysis performed after 18 months of storage at -80°C to assess the long-term impact of freezing on the microbiome
Assess the stability of the microbiome of donor stools after 24months of frozen storage | 24 months of freezing (donor stools)
  Aliquots from a random sample of donations will also be taken for metagenomic analysis performed after 24 months of storage at -80°C to assess the long-term impact of freezing on the microbiome
ESBL-E and CRE infections per 100 patient months at risk (first infection with either) | 6 months
Use of any antibiotics active against all of the colonizing ESBL-E / CRE strains | 6 months
Use of any antibiotics active against at least one of the colonizing ESBL-E / CRE strains | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan J Harbarth, MD, MS, Principal Investigator — Geneva University Hospitals and University of Geneva
Locations (4):
- Assistance Publique-Hôpitaux de Paris, Hôpital Beaujon, Clichy, France
- Sourasky Medical Center, Tel Aviv, Israel
- Universitair Medisch Centrum Utrecht,, Utrecht, Netherlands
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Huttner B, Haustein T, Uckay I, Renzi G, Stewardson A, Schaerrer D, Agostinho A, Andremont A, Schrenzel J, Pittet D, Harbarth S. Decolonization of intestinal carriage of extended-spectrum beta-lactamase-producing Enterobacteriaceae with oral colistin and neomycin: a randomized, double-blind, placebo-controlled trial. J Antimicrob Chemother. 2013 Oct;68(10):2375-82. doi: 10.1093/jac/dkt174. Epub 2013 May 29. PMID 23719234
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Derived] de Lastours V, Poirel L, Huttner B, Harbarth S, Denamur E, Nordmann P. Emergence of colistin-resistant Gram-negative Enterobacterales in the gut of patients receiving oral colistin and neomycin decontamination. J Infect. 2020 May;80(5):578-606. doi: 10.1016/j.jinf.2020.01.003. Epub 2020 Jan 15. No abstract available. PMID 31954100
- [Derived] Huttner BD, de Lastours V, Wassenberg M, Maharshak N, Mauris A, Galperine T, Zanichelli V, Kapel N, Bellanger A, Olearo F, Duval X, Armand-Lefevre L, Carmeli Y, Bonten M, Fantin B, Harbarth S; R-Gnosis WP3 study group. A 5-day course of oral antibiotics followed by faecal transplantation to eradicate carriage of multidrug-resistant Enterobacteriaceae: a randomized clinical trial. Clin Microbiol Infect. 2019 Jul;25(7):830-838. doi: 10.1016/j.cmi.2018.12.009. Epub 2019 Jan 4. PMID 30616014
- See also: Official website of the R-GNOSIS project — http://www.r-gnosis.eu/